CLINICAL TRIAL: NCT01850966
Title: Investigation of the Safety and Efficacy of Iguratimod in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: CRM01T
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis, Rheumatoid, Iguratimod
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — iguratimod

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iguratimod
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — The usual adult dosage for oral use of 25 mg tablet of iguratimod once daily for 4 weeks or more, after which the dosage should be increased to one 25 mg tablet taken twice daily.

SUMMARY:
To investigate the safety and efficacy of the administration of Iguratimod (CRM01T) for 52 weeks in patients with rheumatoid arthritis in clinical practice

ELIGIBILITY:
Inclusion criteria

* Participants with rheumatoid arthritis
* Participants who take iguratimod

Exclusion criteria

* Participants registered for this survey previously
* Pregnant women or women suspected of being pregnant
* Participants with a serious liver disorder
* Participants with peptic ulcer
* Participants with known hypersensitivity to iguratimod or any of its excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals and clinics in Japan
Sampling Method: Non-Probability Sample
Enrollment: 2747 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2014-04-13 (Actual); Study Completion 2014-04-13 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score (DAS28) for Rheumatoid Arthritis (EULAR Response Criteria) | 52 weeks (0-24 weeks and 25-52 weeks)
  DAS28 is a quantitative tool used to measure and monitor disease activity and treatment of rheumatoid arthritis. DAS28 uses a formula that includes the number of tender joints and swollen joints for a maximum of 28 joints.
  DAS28 is used to assess whether an individual participant has a significant improvement of the disease activity, compared to baseline.
  * Good response: Baseline DAS28 less than or equal to 3.2 (low disease activity); DAS28 Improvement >1.2
  * Moderate response: Baseline DAS28 less than or equal to 3.2; DAS28 Improvement >0.6 and less than or equal to 1.2
  * or Baseline DAS28 >3.2 and less than or equal to 5.1; DAS28 Improvement >0.6
  * or Baseline DAS28 >5.1; DAS28 Improvement >1.2
  * No response: Baseline DAS28 >5.1 (high disease activity); DAS28 Improvement less than or equal to 1.2 or DAS28 Improvement less than or equal to 0.6

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Yoshimura, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (453):
- Japan (453):
  - Aisai, Aichi-ken
  - Ama, Aichi-ken
  - Anjo, Aichi-ken
  - Chita, Aichi-ken
  - Gamagōri, Aichi-ken
  - Handa, Aichi-ken
  - Hekinan, Aichi-ken
  - Ichinomiya, Aichi-ken
  - Kasugai, Aichi-ken
  - Kitanagoya, Aichi-ken
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Tokoname, Aichi-ken
  - Toyohashi, Aichi-ken
  - Toyokawa, Aichi-ken
  - Toyota, Aichi-ken
  - Tsushima, Aichi-ken
  - Yatomi, Aichi-ken
  - Minamiakita, Akita
  - Noshiro, Akita
  - Yurihonjō, Akita
  - Hachinohe, Aomori
  - Hirosaki, Aomori
  - Minamitsugaru, Aomori
  - Sannohe, Aomori
  - Abiko, Chiba
  - Awa, Chiba
  - Funabashi, Chiba
  - Hongō, Chiba
  - Ichihara, Chiba
  - Ichikawa, Chiba
  - Kashiwa, Chiba
  - Katori-shi, Chiba
  - Kisarazu, Chiba
  - Matsudo, Chiba
  - Minamibōsō, Chiba
  - Mobara, Chiba
  - Narashino, Chiba
  - Narita, Chiba
  - Sakura, Chiba
  - Sōsa, Chiba
  - Tomisato, Chiba
  - Urayasu, Chiba
  - Yachiyo, Chiba
  - Yotsukaidō, Chiba
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Saijō, Ehime
  - Shikokuchūō, Ehime
  - Uwajima, Ehime
  - Mikatakaminaka, Fukui
  - Sabae, Fukui
  - Tsuruga, Fukui
  - Chikushi, Fukuoka
  - Fukutsu, Fukuoka
  - Itoshima, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Munakata, Fukuoka
  - Nakama, Fukuoka
  - Omuta, Fukuoka
  - Yame, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Iwaki, Fukushima
  - Kōriyama, Fukushima
  - Shirakawa, Fukushima
  - Ibi, Gifu
  - Kakamigahara, Gifu
  - Kamo, Gifu
  - Motosu, Gifu
  - Nakatsugawa, Gifu
  - Ōgaki, Gifu
  - Sekimachi, Gifu
  - Takada, Gifu
  - Agatsuma, Gunma
  - Annaka, Gunma
  - Fujioka, Gunma
  - Isesaki, Gunma
  - Kiryū, Gunma
  - Maebashi, Gunma
  - Ōta, Gunma
  - Shibukawa, Gunma
  - Takasaki, Gunma
  - Aki-takata, Hiroshima
  - Fukuyama, Hiroshima
  - Higashihiroshima, Hiroshima
  - Kure, Hiroshima
  - Onomichi, Hiroshima
  - Takehara, Hiroshima
  - Yamagata, Hiroshima
  - Abashiri, Hokkaido
  - Asahikawa, Hokkaido
  - Bibai, Hokkaido
  - Chitose, Hokkaido
  - Date, Hokkaido
  - Ebetsu, Hokkaido
  - Furano, Hokkaido
  - Hakodate, Hokkaido
  - Honmachi, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Matsumae, Hokkaido
  - Nayoro, Hokkaido
  - Obihiro, Hokkaido
  - Sapporo, Hokkaido
  - Sorachi, Hokkaido
  - Takikawa, Hokkaido
  - Yoichi, Hokkaido
  - Ako, Hyōgo
  - Amagasaki, Hyōgo
  - Ashiya, Hyōgo
  - Himeji, Hyōgo
  - Kako, Hyōgo
  - Katō, Hyōgo
  - Kawanishi, Hyōgo
  - Kobe, Hyōgo
  - Miki, Hyōgo
  - Minamiawaji, Hyōgo
  - Nishinomiya, Hyōgo
  - Ono, Hyōgo
  - Sayō, Hyōgo
  - Sumoto, Hyōgo
  - Takarazuka, Hyōgo
  - Takasago, Hyōgo
  - Tamba, Hyōgo
  - Tatsuno, Hyōgo
  - Chikusei, Ibaraki
  - Higashiibaraki, Ibaraki
  - Hitachi, Ibaraki
  - Hitachi-Naka, Ibaraki
  - Inashiki, Ibaraki
  - Kasama, Ibaraki
  - Kashima-shi, Ibaraki
  - Koga, Ibaraki
  - Mito, Ibaraki
  - Moriya, Ibaraki
  - Ryūgasaki, Ibaraki
  - Toride, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Yūki, Ibaraki
  - Hakui, Ishikawa-ken
  - Kaga, Ishikawa-ken
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Komatsu, Ishikawa-ken
  - Hanamaki, Iwate
  - Ichinoseki, Iwate
  - Kitakami, Iwate
  - Morioka, Iwate
  - Ōfunato, Iwate
  - Ōshū, Iwate
  - Shimohei, Iwate
  - Ayauta, Kagawa-ken
  - Kan’onjichō, Kagawa-ken
  - Marugame, Kagawa-ken
  - Sakaidechō, Kagawa-ken
  - Sanuki, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Akune, Kagoshima-ken
  - Kamikoshikichō-oshima, Kagoshima-ken
  - Kanoya, Kagoshima-ken
  - Soh, Kagoshima-ken
  - Chigasaki, Kanagawa
  - Ebina, Kanagawa
  - Fujisawa, Kanagawa
  - Hiratsuka, Kanagawa
  - Isehara, Kanagawa
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Zushi, Kanagawa
  - Agawa, Kochi
  - Aki, Kochi
  - Kami, Kochi
  - Nankoku, Kochi
  - Shimanto, Kochi
  - Aso, Kumamoto
  - Hitoyoshi, Kumamoto
  - Isshōchi, Kumamoto
  - Minamata, Kumamoto
  - Tamana, Kumamoto
  - Yamaga, Kumamoto
  - Fukuchiyama, Kyoto
  - Jōyō, Kyoto
  - Kameoka, Kyoto
  - Kizugawa, Kyoto
  - Kōtari, Kyoto
  - Kyōtanabe, Kyoto
  - Maizuru, Kyoto
  - Nantan, Kyoto
  - Soraku, Kyoto
  - Uji, Kyoto
  - Yawata, Kyoto
  - Kuwana, Mie-ken
  - Matsusaka, Mie-ken
  - Shima, Mie-ken
  - Suzuka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Higashimatsushima, Miyagi
  - Ishinomaki, Miyagi
  - Iwanuma, Miyagi
  - Kesennuma, Miyagi
  - Murata, Miyagi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Hyūga, Miyazaki
  - Kobayashi, Miyazaki
  - Kushima, Miyazaki
  - Miyakonojō, Miyazaki
  - Saito, Miyazaki
  - Azumino, Nagano
  - Chiisagata, Nagano
  - Hanishina, Nagano
  - Iida, Nagano
  - Iiyama, Nagano
  - Ina, Nagano
  - Kamiminochi, Nagano
  - Komoro, Nagano
  - Matsumoto, Nagano
  - Okaya, Nagano
  - Saku, Nagano
  - Shimoina, Nagano
  - Shiojiri, Nagano
  - Suwa, Nagano
  - Ueda, Nagano
  - Ōmura, Nagasaki
  - Sasebo, Nagasaki
  - Kashiba, Nara
  - Kashihara, Nara
  - Kitakatsuragi, Nara
  - Ōuda-yamaguchi, Nara
  - Shiki, Nara
  - Yamatokōriyama, Nara
  - Yamatotakada, Nara
  - Yoshinoyama, Nara
  - Jōetsu, Niigata
  - Kamo, Niigata
  - Sado, Niigata
  - Sanjō, Niigata
  - Shibata, Niigata
  - Beppu, Oita Prefecture
  - Kunisaki, Oita Prefecture
  - Nakatsu, Oita Prefecture
  - Saiki, Oita Prefecture
  - Yufu, Oita Prefecture
  - Asakuchi, Okayama-ken
  - Kurashiki, Okayama-ken
  - Setouchi, Okayama-ken
  - Tsukubo, Okayama-ken
  - Naha, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Daitō, Osaka
  - Habikino, Osaka
  - Hannan, Osaka
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Ibaraki, Osaka
  - Ikeda, Osaka
  - Izumiōtsu, Osaka
  - Izumisano, Osaka
  - Kadoma, Osaka
  - Kaizuka, Osaka
  - Katano, Osaka
  - Kishiwada, Osaka
  - Mino, Osaka
  - Mishima, Osaka
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Sennan, Osaka
  - Settsu, Osaka
  - Shijōnawate, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Toyonaka, Osaka
  - Ogi, Saga-ken
  - Takeo, Saga-ken
  - Taku, Saga-ken
  - Tosu, Saga-ken
  - Chichibu, Saitama
  - Fujimi, Saitama
  - Fujimino, Saitama
  - Fukaya, Saitama
  - Gyōda, Saitama
  - Hasuda, Saitama
  - Hidaka, Saitama
  - Higashi-Matsuyama, Saitama
  - Hiki, Saitama
  - Iruma, Saitama
  - Kasukabe, Saitama
  - Kawagoe, Saitama
  - Kawaguchi, Saitama
  - Kitakatsushika, Saitama
  - Kitamoto, Saitama
  - Koshigaya, Saitama
  - Kumagaya, Saitama
  - Minamisaitama, Saitama
  - Niiza, Saitama
  - Osato, Saitama
  - Satte, Saitama
  - Sayama, Saitama
  - Sōka, Saitama
  - Tokorozawa, Saitama
  - Tsurugashima, Saitama
  - Wako, Saitama
  - Yashio, Saitama
  - Gamo, Shiga
  - Higashiōmi, Shiga
  - Kōka, Shiga
  - Kusatsu, Shiga
  - Moriyama, Shiga
  - Nagahama, Shiga
  - Ōtsu, Shiga
  - Izumo, Shimane
  - Matsue, Shimane
  - Oda, Shimane
  - Oki, Shimane
  - Yasugi, Shimane
  - Fuji, Shizuoka
  - Fujieda, Shizuoka
  - Gotemba, Shizuoka
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Kamo, Shizuoka
  - Mishima, Shizuoka
  - Numazu, Shizuoka
  - Syuchi, Shizuoka
  - Tagata, Shizuoka
  - Yaizu, Shizuoka
  - Ashikaga, Tochigi
  - Mooka, Tochigi
  - Nasushiobara, Tochigi
  - Nikkō, Tochigi
  - Oyama, Tochigi
  - Ōmiya, Tochigi
  - Sano, Tochigi
  - Shimotsuke, Tochigi
  - Utsunomiya, Tochigi
  - Anan, Tokushima
  - Miyoshi, Tokushima
  - Okuno, Tokushima
  - Yoshinogawa, Tokushima
  - Adachi City, Tokyo
  - Akiruno, Tokyo
  - Akishima, Tokyo
  - Arakawa City, Tokyo
  - Bunkyo, Tokyo
  - Chiyoda City, Tokyo
  - Chōfu, Tokyo
  - Chūō, Tokyo
  - Edogawa City, Tokyo
  - Fuchū, Tokyo
  - Hachiōji, Tokyo
  - Higashikurume, Tokyo
  - Hino, Tokyo
  - Katsushika-ku, Tokyo
  - Kita-ku, Tokyo
  - Koganei, Tokyo
  - Kokubunji, Tokyo
  - Koto, Tokyo
  - Machida, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Mitaka, Tokyo
  - Musashimurayama, Tokyo
  - Musashino, Tokyo
  - Nakano City, Tokyo
  - Nerima City, Tokyo
  - Ōme, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - Suginami, Tokyo
  - Sumida City, Tokyo
  - tabashi City, Tokyo
  - Tachikawa, Tokyo
  - Taitō City, Tokyo
  - Tama, Tokyo
  - Toshima City, Tokyo
  - Kurayoshi, Tottori
  - Sakaiminato, Tottori
  - Tohaku, Tottori
  - Yonago, Tottori
  - Himi, Toyama
  - Imizu, Toyama
  - Kurobe-shi, Toyama
  - Nakaniikawa, Toyama
  - Nanto, Toyama
  - Oyabe, Toyama
  - Shimoniikawa, Toyama
  - Takaoka, Toyama
  - Tonami, Toyama
  - Arida, Wakayama
  - Nishimuro, Wakayama
  - Tanabe, Wakayama
  - Higashimurayama, Yamagata
  - Nishiokitama, Yamagata
  - Shinjō, Yamagata
  - Tendō, Yamagata
  - Tsuruoka, Yamagata
  - Yonezawa, Yamagata
  - Hōfu, Yamaguchi
  - Nagato, Yamaguchi
  - Shimonoseki, Yamaguchi
  - Shūnan, Yamaguchi
  - Ube, Yamaguchi
  - Chūō, Yamanashi
  - Fuefuki, Yamanashi
  - Kai, Yamanashi
  - Kofu, Yamanashi
  - Minamikoma, Yamanashi
  - Nirasaki, Yamanashi
  - Akita
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Miyagi
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nara
  - Niigata
  - Okayama
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokushima
  - Tottori
  - Toyama
  - Wakayama
  - Yamagata
  - Yamaguchi

REFERENCES:
- [Result] Mimori T, Harigai M, Atsumi T, Fujii T, Kuwana M, Matsuno H, Momohara S, Takei S, Tamura N, Takasaki Y, Ikeuchi S, Kushimoto S, Koike T. Safety and effectiveness of 24-week treatment with iguratimod, a new oral disease-modifying antirheumatic drug, for patients with rheumatoid arthritis: interim analysis of a post-marketing surveillance study of 2679 patients in Japan. Mod Rheumatol. 2017 Sep;27(5):755-765. doi: 10.1080/14397595.2016.1265695. Epub 2016 Dec 21. PMID 27919207
- [Result] Rheumatology. 2018;59: 222-32.